CLINICAL TRIAL: NCT05322902
Title: Comparison of Intraoperative Remifentanil Requirements During Remimazolam Versus Propofol Total Intravenous Anesthesia With Analgesia Nociception Index-guided Remifentanil Administration: a Randomized Controlled Study
Brief Title: Remimazolam Total Intravenous Anesthesia Under Analgesia Nociception Index-guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Profeesor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2022-0039
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty; Remimazolam
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Total intravenous anesthesia with remimazolam and remifentanil
  Interventions: Drug: remimazolam group
- Propofol group (Active Comparator): Total intravenous anesthesia with propofol and remifentanil
  Interventions: Drug: propofol group

INTERVENTIONS:
Drug: remimazolam group — Remimazolam 6 mg/kg/hr is administered as an intravenous infusion until the patient loses consciousness. Anesthesia is maintained at 1 mg/kg/hr of remimazolam. After confirming that the eyelash reflex disappears, rocuronium 0.8 mg/kg is administered, and SGA insertion is performed. During maintenance of general anesthesia, the concentration of remifentanil is continuously adjusted so that the ANI is above 50.
  Arms: Remimazolam group
Drug: propofol group — Propofol intravenous infusion is initiated by the application of a target concentration infusion (TCI) pump to cause the patient to lose consciousness. After confirming that the eyelash reflex disappears, rocuronium 0.8 mg/kg is administered, and SGA insertion is performed. During maintenance of general anesthesia, the concentration of remifentanil is continuously adjusted so that the ANI is above 50.
  Arms: Propofol group

SUMMARY:
The investigators hypothesized that intraoperative opioid consumption would be different between remimazolam and propofol if the ANI-guided remifentanil continuous infusion rate was adjusted when the depth of anesthesia was maintained at similar depths with remimazolam or propofol under total intravenous anesthesia. The purpose of this study is to compare the intraoperative remifentanil requirement in patients undergoing total knee arthroplasty when the intraoperative remifentanil dose adjustment was performed under the ANI guidance while maintaining a similar depth of anesthesia with remimazolam or propofol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19~80 years of age who are expected to elective total knee arthroplasty under general anesthesia
2. ASA PS 1-3

Exclusion Criteria:

1. Second total knee arthroplasty under a prior plan of staged total knee arthroplasty, both
2. Previous hepatectomy or liver transplant
3. Estimated glomerular filtration rate < 30 mL/min/1.73m2
4. Patients with moderate or more hepatic impairment (AST/ALT is more than 2.5 times the upper limit of normal)
5. Uncontrolled hypertension (systolic blood pressure > 160mmHg)
6. Acute narrow angle glaucoma
7. Myasthesia gravis
8. Known allergy to the drugs included in the study
9. Cardiac arrhthmia (non-sinus rhythm)
10. Taking drugs that affect the autonomic nervous system of diabetes
11. Psychiatric or neurologic disease (major depression disorder, dementia or cerebral infarction)
12. History of drug or alcohol abuse

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption (mcg/kg/min) | Day 0, intraoperative
  At the start of anesthesia induction, intravenous remifentanil infusion is started and the intraoperative remifentanil infusion rate is adjusted based on the ANI 50 during surgery. The total dose of remifentanil infused intraoperatively is recorded.

SECONDARY OUTCOMES:
Numeric rating scale pain score at rest | up to 24 hours after the surgery
  Pain intensity at rest will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) 1, 6, 24 hours after the surgery.
Postoperative opioid consumption | up to 24 hours after the surgery
  Postoperative opioid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No